CLINICAL TRIAL: NCT03984747
Title: Study for the Prediction of Active Rejection in Organs Using Donor-derived Cell-free DNA Detection
Acronym: SPARO
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-038-TRP
Record Dates: First submitted 2018-11-06; First posted 2019-06-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-04

CONDITIONS: Transplant Rejection; Allograft Rejection; Complications
Keywords: transplant; kidney; renal; allograft; cell-free DNA; lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each participant will provide between 1 to 4 tubes of whole blood (dependent on age) and optional urine collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adult Transplant Patients: Adult subjects who have undergone at least one organ transplant prior to enrollment and are willing to provide consent.
- Pediatric Transplant Patients: Pediatric subjects between ages 2-17 who have undergone at least one organ transplant prior to enrollment and are willing to provide assent/LAR is willing to provide consent.
- Pregnant Transplant Patients: Pregnant subjects who have undergone at least one organ transplant prior to enrollment and are willing to provide consent.

SUMMARY:
This is a multi-center prospective study designed to collect blood samples from transplant patients in order to improve Natera's method for determining allograft rejection status using the donor-derived cell-free DNA analysis, called Prospera.

DETAILED DESCRIPTION:
This is a multi-center prospective study designed to collect blood samples from transplant patients in order to improve Natera's method for determining allograft rejection status using the donor-derived cell-free DNA analysis, called Prospera.

Subjects who have had an organ transplant, who present at the clinic for a standard of care visit or consent for an extra research blood samples to be taken by mobile phlebotomy, meet the study's eligibility criteria and are willing to participate in this research, will be consented and enrolled in this study.

Subjects will provide at least one blood sample at study enrollment and up to three optional follow-up blood samples at future visits. Relevant medical data will also be collected for each patient enrolled.

Urine samples may also be collected at the above described time-points.

Up to 500 subjects over the age of 2 worldwide who meet the study eligibility criteria are expected to be enrolled in this study. The study includes adult, pregnant, and pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 2 years old or older at the time of enrollment
* Subject or Legally Authorized Representative is willing and able to sign the informed consent form (and assent form, if applicable), prior to participation in any study-related procedures.
* Subject has received at least one organ transplant prior to enrollment.

Exclusion Criteria:

* Pediatric subjects under 2 years old
* Subject received donor organ from an identical twin

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As in Inclusion and Exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
To develop an assay to detect allograft rejection status in transplant patients involving amplification of donor-derived cell-free DNA from donor recipient blood. | 1-3 years
  The primary outcome of the assay developed in this study would be allograft rejection high risk or low risk. This assay result will be compared to the biopsy pathology report which assesses if the transplant organ is in a state of rejection, or not. We are also measuring the donor cell free DNA, which is presumably indicating of an organ being rejected or not. Alterations in the cut off of that donor derived cell free DNA level that is allocated to high risk of rejection will be explored. Sensitivity and specificity of our assay will be calculated as needed for the purpose of validating and improving our technology in detecting donor derived cfDNA from a transplant recipient's blood. No results will be reported to patients or their treating physicians.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Natera Inc., San Carlos, California
  - Balboa United California Institute of Renal Research, San Diego, California
  - Children's Hospital at Montefiore, The Bronx, New York
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
12.4.1 All laboratory specimens, evaluation forms, reports, and other records will be handled in a manner designed to maintain research participant confidentiality. All records will be kept in a secure storage area with limited access. Clinical information will not be released without the written permission of the research participant's guardian except as necessary for monitoring and auditing by the Sponsor, its designee, regulatory bodies, or the IRB, or the DSMB.
  12.4.2 The Principal Investigator or Sub-Investigator and all employees and coworkers involved with this study may not disclose or use for any purpose other than performance of the study, any data, record, or other unpublished, confidential information disclosed to those individuals for the purpose of the study. Prior written agreement from the Sponsor or its designee must be obtained for the disclosure of any said confidential information to other parties

REFERENCES:
- [Background] Sigdel TK, Archila FA, Constantin T, Prins SA, Liberto J, Damm I, Towfighi P, Navarro S, Kirkizlar E, Demko ZP, Ryan A, Sigurjonsson S, Sarwal RD, Hseish SC, Chan-On C, Zimmermann B, Billings PR, Moshkevich S, Sarwal MM. Optimizing Detection of Kidney Transplant Injury by Assessment of Donor-Derived Cell-Free DNA via Massively Multiplex PCR. J Clin Med. 2018 Dec 23;8(1):19. doi: 10.3390/jcm8010019. PMID 30583588
- See also: Optimizing Detection of Kidney Transplant Injury by Assessment of Donor-Derived Cell-Free DNA via Massively Multiplex PCR — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6352163/pdf/jcm-08-00019.pdf